CLINICAL TRIAL: NCT05934344
Title: Assessment of Motor and Social Changes Following Intervention With Observation/Action Training (AOT) Among Patients With Mild Cognitive Impairment
Brief Title: Effectiveness of an Intervention Using Observation/Action Therapy Among Patients With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Estrada Barranco, Clinical Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Universidad Europea
Record Dates: First submitted 2023-05-25; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Mild Cognitive Impairment; Age-associated Memory Impairment
Keywords: Action observation treatment; Dementia; Cognitive impairment; Mirror neurons; Elderly people
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observational learning from the therapist (Experimental): Patients with MCI (Mild Cognitive Impairment) will undergo intervention using therapist-led imitation exercises. They will engage in a 5-week exercise program based on observation and action. Data will be collected at the beginning and end of the program.
  Interventions: Other: Action observation training
- peer learning (Experimental): Patients with MCI (Mild Cognitive Impairment) will undergo intervention using exercises by imitation from individuals residing in the facility but without cognitive impairment. They will participate in a 5-week exercise program based on observation and action. Data will be collected at the beginning and end of the program.
  Interventions: Other: Action observation training
- control group (No Intervention): Patients with cognitive impairment who will receive the standard treatment provided by the facility.

INTERVENTIONS:
Other: Action observation training — The activities proposed will be based on items from the FMA scale (Voluntary movement within synergies, voluntary movement mixing synergies, voluntary movement with little or no synergy, grip, coordination/speed, passive joint movement), and the exercises for the lower limbs will be designed by the authors of the study, based on Vivifrail (32), a multicomponent physical training program for the prevention of deconditioning and falls in older adults. These exercises will be progressive each week, focusing on strengthening, balance, and functional exercises to improve gait. The sessions will last between 20 and 30 minutes, with a frequency of three days per week. The intervention will last for 5 weeks.
  Arms: Observational learning from the therapist; peer learning

SUMMARY:
Mild cognitive impairment (MCI) is a transitional state between normal aging and early dementia, characterized by memory deficits without functional impairment. Cognitive decline prevalence is increasing in older adults, impacting independence and quality of life. Motor dysfunctions, often overlooked in MCI, contribute to these limitations. Action Observation Therapy (AOT), a rehabilitation approach involving observing and imitating motor gestures, promotes brain plasticity through the mirror neuron system. While AOT has shown effectiveness in various populations, its application in MCI is understudied. This study aims to investigate the effects of AOT on cognition, upper and lower limb function, daily activities, gait, and balance in MCI patients. It also compares outcomes when patients observe therapists or MCI individuals with similar characteristics. Primary objectives include comparing AOT efficacy between these groups and a control group. Secondary objectives focus on upper limb functionality, daily activities, balance, cognition, and gait.

DETAILED DESCRIPTION:
Introduction The term MCI (Mild Cognitive Impairment) refers to the transitional state between normal cognitive changes associated with aging and very early dementia. It is a disorder characterized by impairments in both short-term and long-term memory, but without functional deficits. MCI is considered a precursor to dementia.

According to the World Health Organization (WHO), it was estimated that in 2014 there were 5.0 million adults with cognitive impairment (CI) in the population aged 65 years and older, and it is projected that by 2060, this number will increase to nearly 14 million. A study by Gómez on sentinel health networks in Spain describes a prevalence of MCI among individuals aged 65 years and older ranging from 14.5% to 17.6% , which increases with age. Another study reports a prevalence of 11.6% in individuals aged 65 to 69 years, which rises to an average of 22.9% among those aged 85 years and older. Furthermore, a meta-analysis of 9 Spanish studies on different types of dementia showed a prevalence ranging from 3.2% to 12.3% in individuals aged 70 years and older, with higher prevalence in women and increasing with age.

Activities of daily living (ADL) rely on a combination of motor, cognitive, and socioemotional skills . Therefore, CI can directly impact independence in ADL, leading to immobility and social isolation . These factors increase the likelihood of individuals with CI requiring admission to specialized care centers.

Gait and balance impairments are common in individuals with dementia, including slower gait speeds, decreased stride length, altered swing time, among others. However, these motor alterations are often overlooked when addressing CI . Balance impairment combined with gait deficits significantly increases the risk of falls, with approximately 60% of individuals with CI experiencing falls annually, twice as frequently as cognitively intact counterparts . Individuals with CI are also more prone to falls resulting in injuries, with up to a three-fold increase in the incidence of hip fractures compared to those without CI. Recognizing and addressing this connection between cognitive and motor deficits is crucial .

A systematic review from 2018 concluded that combining physical training with cognitive training in a functional context can help mitigate some aspects of CI. Therefore, the evidence supports that cognitive intervention should be concurrent with physical exercises rather than separate .

Action Observation Therapy (AOT) involves observing a motor gesture performed by another individual and then imitating the same movement. This technique has been developed as a physical rehabilitation approach that promotes brain plasticity by activating the mirror neuron system . Previous studies have demonstrated the effectiveness of action observation learning. A study conducted with children with cerebral palsy, presented by Naura et al. , showed that motor learning through observation is more effective and provides more evident benefits when subjects learn from other patients with the same condition but less severity, compared to learning by observing a therapist or another person without motor impairment. However, these results have not been corroborated in older patients or those with CI.

The current literature includes various studies consistently demonstrating that AOT is an effective way to learn or improve specific motor skills. Buccino's work summarizes several studies that have employed AOT, including one in which the intervention was carried out with healthy individuals to imitate a motor action in a new environment for them. Another study showed that AOT facilitates motor learning and the construction of a motor memory trace in adults and in patients who have had a stroke. In another study, it was demonstrated that, in healthy adults, AOT is superior to motor imagery as a strategy for learning a complex motor task, at least in the early phase of motor learning. Buccino concludes that these results can have significant implications in educational activities, sports training, and neurorehabilitation.

Specifically in the field of pathology, evidence exists regarding the application of AOT for upper limb rehabilitation in patients who have had a stroke. A pilot study by Yu-Wei Hsieh concluded that AOT resulted in improvements in most outcomes, suggesting it as a promising alternative to contemporary bilateral arm training interventions (i.e., active control intervention) for subacute stroke patients . In a randomized controlled pilot study by Mancuso et al., it was proposed that AOT is a promising treatment for functional recovery and upper limb function in individuals with moderate to severe upper limb impairment following a stroke. AOT could become a useful strategy in stroke rehabilitation programs, as it improves functionality of the paretic upper limb and allows for regaining maximum independence in ADL . Evidence also exists for AOT in children diagnosed with cerebral palsy, specifying that AOT increases spontaneous use of the affected upper limb through observation and imitation of actions, encouraging children to participate in daily activities. By focusing on functional goals or representing everyday activities, these proposed activities promote automatic use within the everyday environment .

However, upon conducting a search for articles and information, no studies on AOT in patients with MCI for upper limb or lower limb activities were found. The closest finding was an article by Rojasavastera, Rommanee et al., in which AOT combined with gait training was used to improve gait and cognition in older adults with MCI. This is why the proposal for this study was initiated (20).

Therefore, the aim of this study is to investigate whether applying AOT in a population with MCI would yield positive results in cognitive status, upper limb function, ADL, gait, and balance. Furthermore, the study aims to determine whether there are better outcomes when AOT is conducted under the guidance of a therapist or under the direction of MCI-free individuals, compared to self-directed AOT.

Hypothesis and Objectives:

The hypothesis of this study is that intervention using an exercise plan for upper and lower limbs through action observation learning is effective in improving cognitive status, functionality, ADL, gait, and balance in patients with mild cognitive impairment. It is also hypothesized that this effectiveness is greater when the learning process involves observing actions performed by other patients with similar characteristics, compared to observing actions performed by the therapist.

Main Objective:

To compare the effectiveness of action observation therapy in patients with mild cognitive impairment who observe the therapist, patients with mild cognitive impairment who observe patients without cognitive impairment, and a control group.

Secondary Objectives:

To assess the benefits of an exercise plan using action observation learning on upper limb functionality.

To evaluate the effectiveness of an exercise plan using action observation learning on ADL in patients.

To examine the benefits of an exercise plan using action observation learning on balance.

To determine the effects of an exercise plan using action observation learning on cognitive status.

To investigate the impact of an exercise plan using action observation learning on gait.

ELIGIBILITY:
Inclusion Criteria:

* Residents or day care center users without visual or auditory impairments that cannot be corrected with the use of devices (such as glasses or hearing aids) and without any conditions affecting their upper limbs.
* Residents with mild cognitive impairment (MoCA score <26) (23).
* Patients capable of walking at least 10 meters without severe pain in the lower limbs (according to the Visual Analog Scale).
* Patiens capable to perform the tests without the use of external aids or with the use of assistive devices such as a cane, and without medical contraindications for exercise.

Exclusion Criteria:

* The patients without cognitive impairment will be selected based on a MoCA score ranging from 26 to 30,
* Patients without any other neurological or musculoskeletal pathology.
* Patients with no upper limb disorders.
* Patients inability to complete the intervention full-time,
* Patients with presence of aggressive behavior or disturbances,
* Patients with inability to communicate verbally.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Changes cognitive impairment | Before and after the intervention: 5 weeks
  Montreal Cognitive Assessment (MoCA)
Changes Activities of daily living | Before and after the intervention: 5 weeks
  Barthel index
Changes Functionality | Before and after the intervention: 5 weeks
  Fugl-meyer scale
Changes Upper limb dexterity | Before and after the intervention: 5 weeks
  Box and block test
Changes balance | Before and after the intervention: 5 weeks
  Berg Balance Scale
Changes gait | Before and after the intervention: 5 weeks
  10 Meters Walking Tes

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Estrada Barranco, PhD, Study Director — Universidad Europea de Madrid
Locations (1):
- Cecilia Estrada Barranco, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No